CLINICAL TRIAL: NCT03065166
Title: Effects of CabernayZyns (Dried Cabernet Grapes) Intake on Vascular Function and Platelet Reactivity in Postmenopausal Women
Brief Title: Dried Cabernet Grapes and Cardiovascular Risk Markers
Acronym: RZN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 944091
Record Dates: First submitted 2017-02-14; First posted 2017-02-27 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Healthy, Postmenopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raisin Treatment (Experimental): 3.2 ounces of dried Cabernet wine grapes.
  Interventions: Other: Raisin Treatment; Other: Bagel Control
- Bagel Control (Other): One 95g whole wheat bagel.
  Interventions: Other: Raisin Treatment; Other: Bagel Control

INTERVENTIONS:
Other: Raisin Treatment — Subjects will consume 3.2oz of dried Cabernet grapes during a single intervention time point.
Other: Bagel Control — Subjects will consume 95g of whole wheat bagel during a single intervention time point.

SUMMARY:
This study assesses the acute effects of dried Cabernet grape intake on vascular function and platelet reactivity in postmenopausal women. Previous studies from this lab and others have demonstrated acute effects on vascular function and platelet reactivity from phenolic-rich food sources. Postmenopausal women are suggested as the study group, as they are likely to have compromised vascular function due to the loss of protective estrogen, and have been the study group for past and present research projects in this lab.

DETAILED DESCRIPTION:
The initiation and progression of atherosclerotic cardiovascular disease (CVD) is multifactorial in nature, and is currently thought of as a chronic inflammatory condition. To reduce the risk of CVD and its associated health care costs in California and elsewhere, nutrition and health recommendations strongly advocate the consumption of a diet rich in fruits and vegetables. Such recommendations are based largely on epidemiological data; the mechanisms underlying the putative positive effects of plant food-rich diets are poorly defined and an area of active debate.

In addition to essential vitamins and minerals, fruits and vegetables contain a number of bioactive compounds that may be involved in vascular function. In this regard, epidemiological studies have noted a significant inverse relationship between the intake of plant foods rich in polyphenols and the risk of both all-cause mortality and CVD. For example, the "French paradox" refers to diet patterns that, despite being high in saturated fat, are associated with a relatively low cardiovascular risk, which may be due, in part, to a robust intake of polyphenols found in red wine, grapes, and other plant foods. Red wine contains an array of phytochemicals that have been proposed to improve cardiovascular health, with a great focus on polyphenols. However, grape products such as dried cabernet grapes also contain substantial amounts of polyphenols that may be vasculoprotective.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female: 50-70 years
* Women: lack of menses for at least one year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 40 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI ≥ 40 kg/m2
* Dislike or allergy for grape products and raisins
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Alcohol consumption > 3 drinks/week (i.e. 1 bottle of beer, 1 glass of wine, and 1 shot of hard liquor)
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day for females
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Use of multi-vitamin and mineral other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL].

(using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);

* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

The following special populations will be excluded:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Postprandial Micro-vascular Function | Baseline and 2-hour measures on day 0 and day 7.
  To determine whether an acute intake of dried Cabernet grapes will improve vascular function, as measured using peripheral artery tonometry (PAT).

SECONDARY OUTCOMES:
Platelet Aggregation | Baseline and 2-hour measures on day 0 and day 7.
  To determine whether an acute intake of dried Cabernet grapes will alter platelet reactivity, as measured by Chrono-log platelet aggregometer device.
Nitrate/Nitrite | Baseline and 2-hour measures on day 0 and day 7.
  Blood analysis to determine whether an acute intake of dried Cabernet grapes will affect plasma circulating nitrate and nitrite levels.
Baseline Complete Metabolic Panel | Baseline measures on day 0 and day 7.
  Blood analyses will include measurements of complete blood cell count, comprehensive metabolic panel, and lipid profile.
Postprandial Complete Metabolic Panel | 2-hour measures on day 0 and day 7.
  Blood analyses will include measurements of complete blood cell count, comprehensive metabolic panel, and lipid profile.
Body Weight | Baseline measure on day 0 and day 7.
  Body weight will be recorded at baseline on initial visit as well as visit one week after.
Blood Pressure | Baseline measure on day 0 and day 7.
  The office blood pressure measurement will be obtained (3 measurements 5 minutes apart after a 15 minute rest).

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No